CLINICAL TRIAL: NCT07274579
Title: Development and Real-World Validation of an Intelligent Interpretation Model for Claudin18.2 Protein Expression in Digestive System Tumors
Brief Title: An Artificial Intelligence Model for Aiding Claudin18.2 Expression Diagnosis in Gastric Adenocarcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Qianfoshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-619
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Digestive Oncology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples Without DNA: Samples retained, with no potential for DNA extraction from any retained samples (e.g., fixed tissue, plasma)

GROUPS / COHORTS (3):
- Prospective validation dataset: We conducted a prospective validation study to compare the diagnostic performance among pathologists, our pathology foundation model, and pathologist-with-AI-assisted diagnosis. This study was initiated on October 1, 2025 at Nanfang Hospital, Southern Medical University (NFHSMU)
- QFSH external validation dataset: 2000 slides from 1000 eligible individuals were obtained in the Qianfoshan Hospital (QFSH, Jinan, China) between January 2020 and February 2026, which was used to validate the model.
- Randomized controlled trial: We conducted a randomized controlled trial（RCT）to compare the diagnostic performance among pathologists, the pathology foundation model, and pathologist-with-model-assisted diagnosis at Nanfang Hospital of Southern Medical University (NFHSMU).The trial commenced data collection on February 1, 2023 to establish the NFHSMU randomized controlled trial dataset. Following quality control, the slides were randomly allocated (1:1 ratio) into three groups:Pathologist-only group/Model-assisted pathologist group.

SUMMARY:
The investigators plan to develop a deep learning-based automatic interpretation model for Claudin18.2(CLDN18.2) using the institution's and multiple other centers' extensive pathological resources of digestive system adenocarcinomas. This study will not only strictly follow the latest domestic expert consensus and standards, but also aims to address current pain points in manual interpretation. It seeks to provide technical support for standardizing, objectifying, and streamlining CLDN18.2 testing, thereby advancing the application of precision medicine in the diagnosis and treatment of digestive system diseases. The project has clear clinical necessity and broad application prospects.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years.
2. Patients who underwent CLDN18.2 immunohistochemistry and H&E staining.
3. Availability of complete pathology reports and clinical information.

Exclusion Criteria:

1.Patients with missing data or specimens not meeting quality control requirements for analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inclusion criteria comprised patients aged over 18 years with definitive pathological diagnoses.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve (AUC) | Diagnostic evaluation will be performed within 1 week when the whole slide images(WSIs) are obtained.
  Area under the curve

SECONDARY OUTCOMES:
Specificity | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  The true negative rate (TNR) of the diagnostic platform, which is the ratio between the number of negative individuals correctly categorized by platform and the total number of actual negative individuals (%).
Sensitivity | Diagnostic evaluation will be performed within 1 week when the WSIs are obtained
  The true positive rate (TPR) of the diagnostic platform, which is the ratio between the number of positive individuals correctly categorized by platform and the total number of actual positive individuals (%).

CONTACTS AND LOCATIONS:
Overall Officials: Li Liang, Study Director — Nanfang Hospital, Southern Medical University
Locations (2):
- China (2):
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - Qianfoshan Hospital, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No
Requests for the data collected and analyzed in this study will be considered if the application is in line with public benefits and the applicant is willing to sign a data access agreement. Contact can be through the corresponding author.